CLINICAL TRIAL: NCT06818890
Title: Comparison of the Stability of the Peri-implant Hard and Soft Tissues with the Use of One-time Definitive Abutment (on 1 Concept) and the Conventional 2 Stage Implant Connection
Brief Title: Response of Hard and Soft Tissue Around the Dental Implant to 2-Piece Abutment Vs Conventional Restorative Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Sarfaraz (Other)
Collaborators: Yenepoya Dental College (Other)
Responsible Party: Sponsor-Investigator, Hasan Sarfaraz, Professor, Yenepoya Dental College
Organization: Yenepoya Dental College (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018/193
Record Dates: First submitted 2025-02-03; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Partially Edentulous Mandible; Dental Implant; Soft Tissue Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Definite abutment base (Experimental): The On1 base (height 1.75 mm) and the On1 healing cap and On1 abutment (Nobel Biocare AB). it is a two-piece abutment of which the base is connected to the implant on the day of implant placement.
  Interventions: Device: Definitive abutment base
- Conventional healing abutment (Active Comparator): Universal healing abutment and the universal base abutment
  Interventions: Device: Conventional Healing Abutment

INTERVENTIONS:
Device: Definitive abutment base — Definite abutment base, this is a two-piece definitive abutment where the base is connected to the implant as soon as it is placed.This abutment will allow the tissues around the implant to heal undisturbed, thus, establishing a good and healthy periimplant soft and hard tissue with long-term stability.
  Arms: Definite abutment base
Device: Conventional Healing Abutment — A healing abutment of different diameters (4.3, 5, 6 mm) and heights (1.5, 3 mm) is placed on the day of the surgery, and the flaps are sutured around them to allow for tissue healing around the abutment to create an optimum emergence profile and tissue cuff around the implant and definitive abutment.
  Arms: Conventional healing abutment

SUMMARY:
The goal of the study is to determine whether using a two-piece definitive abutment, as opposed to a traditional two-stage healing abutment connection, will reduce the loss of crestal bone surrounding the implant and improve soft tissue adaption. With the use of a manual periodontal probe, it will be recorded at four locations per implant. In order to prevent its removal during healing, an abutment base of the definitive restorative abutment will be positioned during implant surgery. Therefore, there is no departure from the standard course of treatment. An implant and crown will be used to replace a lost tooth, which will benefit the patients.

Benefit to society: more predictable and enhanced functional and aesthetic treatment outcomes.

Benefit to Scientific Advancement: This concept will be beneficial in maintaining the peri-implant soft tissue and bone levels.

Changes in interproximal bone levels will be measured in standardized periapical digital radiographs (x-rays) once a month, which is usually not associated with any complications.

The number of visits to the hospital: On the day of implant placement, 12th-week Impression Visit, 16th-week Prosthesis Placement, 20th-week 1st Month post prosthesis, follow up, 28th-week 3rd-month post prosthesis follow-up, 40th-week 6th-month post prosthesis follow-up, 64th-week 1-year follow-up after placing the definitive restoration. On every visit, radiographs will be taken. Patients should maintain regular oral hygiene to prevent future bone loss.

No one else shall be privy to participants' details. Implant treatment for the participant is free. The participant will give consent for any advisable and necessary dental procedures, medications, or anaesthetics to be administered by the attending dentist or his supervised staff for diagnostic purposes or for implant placement. Also give consent to make radiographic and photographic records; these records may also include study models, x-rays, and blood studies. If implants fail, then they will be retreated free of charge. Participants understood and acknowledged that they agreed to be part of this clinical study, will keep up with the follow-up appointments, and if they want, they can choose to drop out of the study anytime on the course of study. That there is no force or influence to participate, that he/she can take enough time to decide whether to participate, and that he/she can ask any doubts to the PI at any point in time.

DETAILED DESCRIPTION:
An in-vivo clinical assessment and radiologic study protocol was developed and approved by the ethics committee of the Yenepoya University in Mangalore, in accordance with the Declaration of Helsinki. All patients provided written informed consent prior to the performance of any study procedures, and only data collected after the patients had signed informed consent were considered during the study analysis. A single-center, open, randomized parallel-group trial was conducted to compare the peri-implant tissue response of the abutment base treatment (test group) to that of a conventional restorative workflow with a healing abutment (control group). Patients underwent clinical assessments for the replacement of one or more missing mandibular posterior teeth with an implant-supported crown. Pre-operative CBCT scans were taken for all the patients to assess the quality and quantity of bone at the implant recipient sites.

All the surgeries were carried out by a skilled surgeon with minimal hard and soft tissue trauma during which NobelParallel TiUnite CC Implants (Nobel Biocare AB, Göteborg, Sweden) with diameters ranging from 4.3 mm to 5 mm and lengths from 10 mm to 11.5 mm were placed in healed edentulous sites in the posterior mandible in an equicrestal position. All procedures were performed using crestal incision with a full-thickness flap raised. The implants were placed at the crest of alveolar bone; no bone mill was used during the On1 base seating. The patients received broad-spectrum antibiotics for 5 days and analgesics for 2 days. The implant placement (IP) surgery was considered the baseline and was referred to as such. The On1 base (height 1.75 mm) and the On1 healing cap (Nobel Biocare AB) were placed in the test group, while the healing abutment (Conical Connection RP ø 6 x 5 mm; Nobel Biocare AB) was placed in the control group. The soft tissue was sutured (with sutures removed after 1 week), and the site was allowed a 12-week non-submerged healing, at which point the conventional tray impression was taken. At 16 weeks, a prosthetic crown (made in the university lab) was delivered, which was designated as the definitive prosthesis delivery (DPP), The follow-up appointments took place at 1-3-6 months and 1-year post-DPP.

ELIGIBILITY:
Inclusion Criteria:

* Adequate width and height of bone for the placement of appropriate size implant(s).
* Well-healed edentulous sites with a minimum of 2 mm of soft tissue thickness.
* Patients willing to participate by giving informed consent.
* Patients agreeing to attend the planned follow-up visits.

Exclusion Criteria:

* Medically compromised patients where surgery was contraindicated.
* Patients with poor oral hygiene and/or suffering from periodontal disease.
* Patients with insufficient quantity/quality of bone.
* Patient with edentulous sites with a lack of attached gingiva.
* Patients with edentulous sites with insufficient prosthetic space.
* Patients with a history of parafunctional occlusal habits.
* Tobacco or alcohol use or drug dependency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Crestal Bone levels | I year follow up
  The crestal bone level changes at the mesial and distal interproximal areas were captured at baseline (implant placement), 1-, 3-, 6 months, and 1-year post-restoration. Intra-oral periapical digital radiographs using the digital radiograph sensor (Gendex Dental Systems, Kavo, USA) and measured in millimeters using the measuring tool in the bundled software VixWin. The process was standardized by a positioning/paralleling device (Gendex, Kavo, Germany). The radiographs were verified for any distortion by measuring the distance between the head of the implant and the apex and using the known length of the implant. The mesial and distal crestal bone levels were calculated by determining the distance from the implant head to the ﬁrst visible bone contact in millimeters.

SECONDARY OUTCOMES:
Peri-Implant Tissue Health | I year follow up
  A clinical peri-implant soft tissue health assessment was made using four different indices or measures; a positive finding in any of the two indices or measures would indicate compromised tissue health. It was recorded at 2 buccal and 2 lingual sites per implant with the aid of a manual periodontal probe at 4 time intervals: Day of Prosthesis Placement, 1-, 3-, 6-month, and 1-year post prosthesis placement. It was done using modiﬁed plaque index (mPLI with score 0-plaque seen to 3-visibly detectable plaque), modified sulcus bleeding index (mSBI with score 0-no bleeding to 3-heavy or profuse bleeding), mean probing depth (mPD) measured in millimeters with a plastic, color-coded periodontal probe (Mombelli et al. 1987) from 4 different sides: mesiobuccal, distobuccal, mesiolingual, and distolingual, and the width of peri-implant keratinized mucosa (KM) measured in millimeters in the mid-buccal and lingual sites.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Sarfaraz, MDS, Principal Investigator — Yenepoya Dental College
Locations (1):
- Yenepoya Dental College Hospital, Mangaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
As a requirement for ethical clearance, we had informed the patient that their individual data will be kept confidential and will not be shared.